CLINICAL TRIAL: NCT02662257
Title: Impact of Inhalational Versus Intravenous Anesthesia Maintenance Methods on Incidence of Postoperative Delirium in Elderly Patients After Cancer Surgery: An Open-label, Randomized Controlled Trial
Brief Title: Impact of Anesthesia Maintenance Methods on Incidence of Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); The People's Hospital of Ningxia (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Guizhou Provincial People's Hospital (Other); Affiliated Hospital of Qinghai University (Other); The Third Xiangya Hospital of Central South University (Other); Cancer Hospital of Guangxi Medical University (Other); Shanxi Provincial People's Hospital (Other Government); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tang-Du Hospital (Other); Tianjin Nankai Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015[869]-1; ChiCTR-IPR-15006209 (Registry Identifier: Chinese Clincial Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2016-01-05; First posted 2016-01-25 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Delirium; Postoperative Complications; Postoperative Cognitive Dysfunction
Keywords: Sevoflurane; Propofol; Aged; Neoplasm; Surgical Procedure, Operative; Delirium; Postoperative Complications; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Postoperative Complications; Postoperative Cognitive Complications; Neoplasms | interventions — Sevoflurane; Inhalation; Propofol; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sevoflurane group (Active Comparator): Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, sevoflurane inhalational concentration will be decreased and fentanyl/sufentanil will be administered when necessary. Sevoflurane inhalation will be stopped at the end of surgery.
  Interventions: Drug: Sevoflurane
- Propofol group (Experimental): Propofol will be administered by intravenous infusion for anesthesia maintenance. The infusion rate of propofol will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, propofol infusion rate will be decreased and fentanyl/sufentanil will be administered when necessary. Propofol infusion will be stopped at the end of surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, sevoflurane inhalational concentration will be decreased and fentanyl/sufentanil will be administered when necessary. Sevoflurane inhalation will be stopped at the end of surgery.
  Other Names: Sevoflurane for inhalation
  Arms: Sevoflurane group
Drug: Propofol — Propofol will be administered by intravenous infusion for anesthesia maintenance. The infusion rate of propofol will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, propofol infusion rate will be decreased and fentanyl/sufentanil will be administered when necessary. Propofol infusion will be stopped at the end of surgery.
  Other Names: Propofol for injection
  Arms: Propofol group

SUMMARY:
Surgery is one of the major treatment methods for patients with malignant tumor. And, alone with ageing process, more and more elderly patients undergo surgery for malignant tumor. Evidence emerges that choice of anesthetics, i.e., either inhalational or intravenous anesthetics, may influence the outcome of elderly patients undergoing cancer surgery. Delirium is a commonly occurred early postoperative cognitive complication in the elderly, and its occurrence is associated with the worsening outcomes. Choice anesthetics may influence the occurrence of postoperative delirium. However, evidence in this aspect is conflicting.

DETAILED DESCRIPTION:
It is estimated that 234.2 million major surgical procedures are undertaken every year worldwide. Surgery is one of the major treatment methods for patients with malignant tumor. And, alone with ageing process, more and more elderly patients undergo surgery for malignant tumor. Evidence emerges that choice of anesthetics, i.e., either inhalational or intravenous anesthetics, may influence the outcome of elderly patients undergoing cancer surgery.

Delirium is a commonly occurred cognitive complication in elderly patients after surgery. The occurrence of delirium is associated with the worsening outcomes, including increased morbidity and mortality, prolonged hospital stay, elevated medical care cost, and declined cognitive function. High age, major surgery, and critical illness are major risk factors of postoperative delirium (POD). However, the relationship between use of general anesthetics and occurrence of delirium cannot be excluded.

There are studies that compared the effects of two kinds of anesthetics on the cognitive outcomes after surgery. In the study of Nishikawa et al., 50 elderly (≥ 65 years) patients undergoing long-duration laparoscope-assisted surgery randomly received sevoflurane or propofol anesthesia. The results showed that, although the incidence of POD was not significantly different between the two groups, the delirium rating scale (DRS) score was significantly lower in the sevoflurane group than in the propofol group at postoperative days 2-3 (P = 0.007 and 0.002, respectively). In the study of Schoen et al., 128 patients undergoing on-pump cardiac surgery were randomized into two groups. The results showed that early postoperative cognitive function was significantly better in sevoflurane group than in the propofol group, especially in those who experienced cerebral desaturation during surgery.

On the other hand, some studies reported contrary results. In a large sample size study of 2000 patients undergoing general anesthesia, patients carrying ApoE4 epsilon 4 allele were more likely to develop early postoperative cognitive decline after inhalational anesthesia (odd ratio 3.31, 95% confidence interval 1.25-6.39, P < 0.05), but not after intravenous anesthesia (odd ratio 0.93, 95% confidence interval 0.37-2.39, P > 0.05). In a randomized control trail of 44 patients undergoing carotid endarterectomy, the mini-mental state examination (MMSE) score was significantly higher, whereas blood S100B concentration was significantly lower in the propofol group than in the sevoflurane group at 24 hours after surgery. In the study of Tang et al., 200 elderly (≥ 60 years) patients with mild cognitive impairment who planned to undergo radical rectal resection randomly received either sevoflurane or propofol anesthesia. The results showed that, although there was no difference in the incidence of cognitive dysfunction at 7 days after surgery, the negative cognitive effects was more severe after sevoflurane anesthesia than after propofol anesthesia (P = 0.01).

It seems that more evidence suggests the harmful cognitive effects of inhalational anesthetics. However, care must be taken when explaining these results: (1) target patients population were different; (2) sample size were small in the majority of studies; (3) the diagnostic criteria of cognitive complications were different, make it hard to do meta-analysis; (4) the clinical significance the of early postoperative cognitive complication remains to be elucidated.

ELIGIBILITY:
Inclusion criteria

Participants will be included if they meet all the following criteria:

1. Age ≥ 65 years and < 90 years;
2. Primary malignant tumor;
3. Do not receive radiation therapy or chemotherapy before surgery;
4. Scheduled to undergo surgery for the treatment of tumors, with an expected duration of 2 hours or more, under general anesthesia;
5. Agree to participate, and give signed written informed consent.

Exclusion criteria

Patients will be excluded if they meet any of the following criteria:

1. Preoperative history of schizophrenia, epilepsy, parkinsonism or myasthenia gravis;
2. Inability to communicate in the preoperative period (coma, profound dementia, language barrier, or end-stage disease);
3. Critical illness (preoperative American Society of Anesthesiologists physical status classification ≥ IV), severe hepatic dysfunction (Child-Pugh class C), or severe renal dysfunction (undergoing dialysis before surgery);
4. Neurosurgery;
5. Other reasons that are considered unsuitable for participation by the responsible surgeons or investigators (reasons must be recorded in the case report form).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium within 7 days after surgery. | Up to 7 days after surgery
  Delirium is assessed twice daily (8-10 AM and 6-8 PM) with the Confusion Assessment Method for patients without endotracheal intubation or the Confusion Assessment Method for the Intensive Care Unit for patients with endotracheal intubation.

SECONDARY OUTCOMES:
Percentage of intensive care unit (ICU) admission after surgery. | Within 24 hours after surgery.
  Percentage of intensive care unit (ICU) admission after surgery.
Percentage of ICU admission with endotracheal intubation after surgery. | Within 24 hours after surgery.
  Percentage of ICU admission with endotracheal intubation after surgery.
Length of stay in ICU after surgery. | Up to 30 days after surgery.
  Length of stay in ICU after surgery (in patients admitted to the ICU after surgery).
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of non-delirium complications within 30 days. | Up to 30 days after surgery.
  Non-delirium complications are defined as newly occurred events other than delirium that are harmful to patients' recovery and required therapeutic intervention, i.e., grade 2 or higher on the Clavien-Dindo classification.
Cognitive function at 30 days after surgery. | On the 30th day after surgery.
  Cognitive function assessed with Telephone Interview for Cognitive Status-Modified (TICS-m).

OTHER OUTCOMES:
Intensity of pain within 3 days after surgery. | Up to 3 days after surgery.
  Intensity of pain is assessed twice daily (8-10 AM and 6-8 PM) with the Numeric Rating Scale (an 11-point rating scale where 0 = no pain and 10 = the worst pain).
Subjective sleep quality within 7 days after surgery. | Up to 7 days after surgery.
  Subjective sleep quality is assessed once daily (8-10 AM) with the Numeric Rating Scale (an 11-point rating scale where 0 = the worst sleep and 10 = the best sleep).
Cognitive dysfunction assessment | The day before surgery and on the 7th day after surgery
  Cognitive function assessed with a battery of neuropsychological tests before surgery and on the 7th day after surgery. Performed in part of enrolled patients and in control subjects.
Serum vitamine D concentration | The day before surgery
  Blood samples are taken the day before surgery. Serum 25-hydroxyvitamin D concentration is measured with liquid chromatography-mass spectrometry. Performed in part of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (17):
- China (17):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Shenzhen Second People's Hospital, Shenzhen, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hebei Medical University Forth Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital, Nanjing, Jiangsu
  - Ningxia People's Hospital, Yinchuan, Ningxia
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Tang-Du Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Nankai Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Nishikawa K, Nakayama M, Omote K, Namiki A. Recovery characteristics and post-operative delirium after long-duration laparoscope-assisted surgery in elderly patients: propofol-based vs. sevoflurane-based anesthesia. Acta Anaesthesiol Scand. 2004 Feb;48(2):162-8. doi: 10.1111/j.0001-5172.2004.00264.x. PMID 14995937
- [Background] Schoen J, Husemann L, Tiemeyer C, Lueloh A, Sedemund-Adib B, Berger KU, Hueppe M, Heringlake M. Cognitive function after sevoflurane- vs propofol-based anaesthesia for on-pump cardiac surgery: a randomized controlled trial. Br J Anaesth. 2011 Jun;106(6):840-50. doi: 10.1093/bja/aer091. Epub 2011 Apr 25. PMID 21518736
- [Background] Cai Y, Hu H, Liu P, Feng G, Dong W, Yu B, Zhu Y, Song J, Zhao M. Association between the apolipoprotein E4 and postoperative cognitive dysfunction in elderly patients undergoing intravenous anesthesia and inhalation anesthesia. Anesthesiology. 2012 Jan;116(1):84-93. doi: 10.1097/ALN.0b013e31823da7a2. PMID 22108393
- [Background] Kalimeris K, Kouni S, Kostopanagiotou G, Nomikos T, Fragopoulou E, Kakisis J, Vasdekis S, Matsota P, Pandazi A. Cognitive function and oxidative stress after carotid endarterectomy: comparison of propofol to sevoflurane anesthesia. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1246-52. doi: 10.1053/j.jvca.2012.12.009. Epub 2013 May 30. PMID 23725684
- [Background] Tang N, Ou C, Liu Y, Zuo Y, Bai Y. Effect of inhalational anaesthetic on postoperative cognitive dysfunction following radical rectal resection in elderly patients with mild cognitive impairment. J Int Med Res. 2014 Dec;42(6):1252-61. doi: 10.1177/0300060514549781. Epub 2014 Oct 22. PMID 25339455
- [Derived] Cao SJ, Zhang Y, Zhang YX, Zhao W, Pan LH, Sun XD, Jia Z, Ouyang W, Ye QS, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yu JB, Liu ZH, Yin N, Li XY, Ma JH, Li HJ, Wang MR, Sessler DI, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Delirium in older patients given propofol or sevoflurane anaesthesia for major cancer surgery: a multicentre randomised trial. Br J Anaesth. 2023 Aug;131(2):253-265. doi: 10.1016/j.bja.2023.04.024. Epub 2023 Jun 4. PMID 37474241
- [Derived] Zhang Y, Shan GJ, Zhang YX, Cao SJ, Zhu SN, Li HJ, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) Investigators. Preoperative vitamin D deficiency increases the risk of postoperative cognitive dysfunction: a predefined exploratory sub-analysis. Acta Anaesthesiol Scand. 2018 Aug;62(7):924-935. doi: 10.1111/aas.13116. Epub 2018 Mar 26. PMID 29578249
- [Derived] Zhang Y, Li HJ, Wang DX, Jia HQ, Sun XD, Pan LH, Ye QS, Ouyang W, Jia Z, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yang XD, Zhang QG, Yin N, Tan HY, Liu ZH, Yu JB, Ma D. Impact of inhalational versus intravenous anaesthesia on early delirium and long-term survival in elderly patients after cancer surgery: study protocol of a multicentre, open-label, and randomised controlled trial. BMJ Open. 2017 Nov 28;7(11):e018607. doi: 10.1136/bmjopen-2017-018607. PMID 29187413